CLINICAL TRIAL: NCT06993311
Title: Four-year Outcomes of Minimally Invasive XEN Gel Stent Implantation in Pseudoexfoliation Glaucoma: Real World Evidence
Brief Title: Real World Evidence of Xen45 Gel Implant in Pseudoexfoliation Glaucoma
Status: Completed | Type: Observational
Sponsor: Xerencia de Xestión Integrada de Ferrol (Other)
Collaborators: University Hospital Complex of Santiago de Compostela (Unknown)
Responsible Party: Principal Investigator, SARA POSE BAZARRA, Ophthalmologist MD, Xerencia de Xestión Integrada de Ferrol
Other Study IDs: XENPXF
Record Dates: First submitted 2024-05-31; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Pseudoexfoliation Syndrome; Pseudoexfoliation Glaucoma in Both Eyes; Open Angle Glaucoma
Keywords: Xen
MeSH Terms: conditions — Exfoliation Syndrome; Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pseudoexfoliation glaucoma
  Interventions: Device: Xen Gel Stent implantation
- Open-angle glaucoma
  Interventions: Device: Xen Gel Stent implantation

INTERVENTIONS:
Device: Xen Gel Stent implantation — Consecutive patients who underwent either stand-alone Xen stent insertion with MMC(mitomycin C) or combined phacoemulsification between 2018 and 2022

SUMMARY:
The Xen implant is an ab interno device that has been shown to be effective in reducing intraocular pressure in several types of glaucoma, although the evidence in pseudoexfoliative glaucoma is limited. The present retrospective observational study aims to increase knowledge about the long-term effectiveness and safety of the implant in pseudoexfoliative glaucoma. Researchers will compare the results with data from patients with open-angle glaucoma.

ELIGIBILITY:
Inclusion Criteria:

Data will be collected for all patients with pseudoexfoliation glaucoma (PXFG), ocular hypertension (OHT) and pseudoexfoliation syndrome, POAG and other secondary open angle glaucoma (OAG) diagnosed, who underwent surgery from 2018 to 2022.

Patients should be candidates for filtering glaucoma surgery for the following indications:

* uncontrolled intraocular pressure (IOP)
* intolerance or non-adherence to topical treatment
* glaucoma progression despite topical therapy
* surgical cataract patients undergoing phacoemulsification, who were treated with two or more hypotensive drugs and wished to withdraw the medication due to side effects and/or discomfort of the treatment.

Refractory glaucoma and eyes with previous filtering surgery, previous laser treatments or micropulse transscleral cyclophotocoagulation will be also included.

Exclusion Criteria:

* Patients with follow up less than 12 months.
* Patients with end-stage glaucoma, uveitic and angle closure glaucoma.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Data will be collected for all patients with PXFG, POAG and other secondary OAG, who underwent surgery from 2018 to 2022, at 2 terciary care academic ophthalmology centers (University Hospital Complex of Ferrol and University Hospital Complex of Santiago de Compostela, Spain) by 10 surgeons.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
INTRAOCULAR PRESSURE | 12-48 months
  The primary outcome measure will be intraocular pressure reduction at final follow up

SECONDARY OUTCOMES:
NUMBER OF TREATMENTS | 12-48 months
  Number of glaucoma drugs: Investigate the reduction of drugs after surgery
BEST CORRECTED VISUAL ACUITY | 12-48 months
  Best-corrected visual acuity (BCVA): investigators will compare the change of visual acuities (VA) between pre-surgery to last follow-up
RETINAL NERVE FIBER LAYER | 12-48 months
  Retinal nerve fiber layer (RNFL) thickness by optical coherence tomography (OCT): investigators will compare the reduction in the retinal nerve fiber layer by OCT according to the analysis of glaucoma (Heidelberg)
RATES OF REINTERVENTION | 12-48 months
  Number of trabeculectomy or filtering surgery required as a result of poor control of IOP
INCIDENCE OF TREATMENT ADVERSE EVENTS | 12-48 months
  Investigators will determine the safety profile of the intervention through an evaluation of intraoperative and post-operative complications. All adverse events or complications related to the intervention will be recorded in a descriptive manner.
PRESERVATIVES EXPOSURE | 12-48 months
  Investigators will collect data on pre-surgery treatment regarding the use or non-use of preservatives and their exposure time to these drugs to compare effectiveness outcomes in both groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Sara Pose-Bazarra, Ferrol, Spain

IPD SHARING:
Plan to Share IPD: No